CLINICAL TRIAL: NCT04017429
Title: Treatment of Grade III Furcation Defects in Teeth With Low Interproximal Crestal Bone Height, With and Without Osteoplasty, in Conjunction With Open Flap Debridement
Brief Title: Osteoplasty in Conjunction With Surgical Treatment of Mandibular Grade III Furcation Defects (FURC-III-OST)
Acronym: FURC-III-OST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible to recruit and follow-up subjects due to the pandemic
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Anders Verket, Associate Professor, PhD, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FURC-III-OST
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Furcation Defects; Periodontal Diseases
MeSH Terms: conditions — Furcation Defects; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open flap debridement with osteoplasty (Experimental): In this arm, periodontal surgery consists of open flap debridement followed by osteoplasty in the furcation entrance area.
  Interventions: Procedure: Open flap debridement with osteoplasty; Procedure: Open flap debridement without osteoplasty
- Open flap debridement without osteoplasty (Active Comparator): In this arm, periodontal surgery consists of open flap debridement only. No osteoplasty will be performed.
  Interventions: Procedure: Open flap debridement with osteoplasty; Procedure: Open flap debridement without osteoplasty

INTERVENTIONS:
Procedure: Open flap debridement with osteoplasty — Treatment of furcation grade III defect with open flap debridement followed by osteoplasty treatment. Osteoplasty includes altering the bone buccal to the furcation opening to >90 degrees relative to the apico-coronal axis of the tooth.
Procedure: Open flap debridement without osteoplasty — Treatment of furcation grade III defect with open flap debridement only.

SUMMARY:
Teeth with furcation grade III defects will be treated with open flap debridement, with or without osteoplasty. The study is designed to examine the effect of osteoplasty in the treatment of teeth with furcation grade III defects with open flap debridement.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal disease stage III or IV according to 2018 criteria
* Undergoing periodontal therapy (active or supportive) and present 1 or more pair of bilateral mandibular molars affected by furcation involvement grade III with PPD>4mm, and the furcation fornix must be above a tangential line from the distal to mesial interproximal crestal bone level on bitewing radiographs
* Competent to give consent

Exclusion Criteria:

* Previous radiotherapy to the jaws, current use of chemotherapy, systemic long-term corticosteroid treatment
* Present or past use of bisphosphonate treatment
* Pregnant or nursing subjects
* Patients classified as > class II according to ASA classification
* Previous surgical therapy of included furcation defects
* Inhability to comprehend and respond to the quality of life questionnaire
* Dental restorations or prosthesis involving the furcation area
* Root fractures or suspected fractures/infractions
* Caries lesoins in the furcation area
* No systemic antibiotic treatment within 3 months prior to intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Sites with no signs of inflammation | 12 months after treatment
  Proportion of sites without inflammation, defined as no BoP or PPD>4mm following treatment
Sites with no signs of inflammation | 24 months after treatment
  Proportion of sites without inflammation, defined as no BoP or PPD>4mm following treatment

SECONDARY OUTCOMES:
Changes in patient-reported quality of life (QoL) | Preoperatively compared to 24 months after treatment
  To assess QoL changes related to mouth and teeth prior to therapy to after therapy by the use of "The Oral Impacts on Daily Performance (OIDP)" instrument. Each question is assessed by a 5-point scale; (1) never affected; (2) less than once a month; (3) once or twice a month; (4) once or twice a week; and (5) every or nearly every day. The higher number represents more severe impact on quality of life; e.g. worse outcome.
  Each item will be dichotomised yielding the categories (A) affected; including scale categories (2)-(5), and (B) unaffected; including category (1)
Changes in patient-reported quality of life (QoL) | Preoperatively compared to 12 months after treatment
  To assess QoL changes related to mouth and teeth prior to therapy to after therapy by the use of "The Oral Impacts on Daily Performance (OIDP)" instrument. Each question is assessed by a 5-point scale; (1) never affected; (2) less than once a month; (3) once or twice a month; (4) once or twice a week; and (5) every or nearly every day. The higher number represents more severe impact on quality of life; e.g. worse outcome.
  Each item will be dichotomised yielding the categories (A) affected; including scale categories (2)-(5), and (B) unaffected; including category (1)
Loss of clinical attachment level | 12 months after treatment
  To assess further loss of clinical attachment level by the use of a periodontal probe
Loss of clinical attachment level | 24 months after treatment
  To assess further loss of clinical attachment level by the use of a periodontal probe
Number of participants with caries lesions | 24 months after treatment
  To assess caries lesions in furcation defects following therapy. Caries lesions are assessed clinically with an explorer as caries (Y/N)
Radiographic changes | 12 months after treatment
  To assess bone loss as measured on standardized radiographs (in mm)
Radiographic changes | 24 months after treatment
  To assess bone loss as measured on standardized radiographs (in mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Clinical Dentistry, University of Oslo, Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No